CLINICAL TRIAL: NCT01649271
Title: Phase I Trial of Afatinib in Combination With 3 Weekly Trastuzumab in Patients With Tumours Overexpressing HER2. Once the MTD of Afatinib With 3 Weekly Trastuzumab Was Established the Safety of This Dose Will be Assessed Also in Combination With Weekly Trastuzumab.
Brief Title: Phase I Trial of Afatinib and Trastuzumab in HER2 Overexpressing Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.134; 2012-001753-10 (EudraCT Number)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Breast Neoplasms; Stomach Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — Trastuzumab; Afatinib

ARMS (3):
- Phase Ia, group 1 (Experimental): afatinib escalating dose with 3-weekly trastuzumab
  Interventions: Drug: Herceptin; Drug: afatinib
- Phase Ia, group 2 (Experimental): afatinib at MTD dose with weekly trastuzumab
  Interventions: Drug: afatinib; Drug: Herceptin
- Phase Ib (Experimental): afatinib at MTD level with 3-weekly trastuzumab
  Interventions: Drug: trastuzumab; Drug: afatinib

INTERVENTIONS:
Drug: Herceptin — 3-weekly
  Arms: Phase Ia, group 1
Drug: afatinib — at MTD level
  Arms: Phase Ia, group 2
Drug: trastuzumab — 3-weekly
  Arms: Phase Ib
Drug: Herceptin — weekly
  Arms: Phase Ia, group 2
Drug: afatinib — at MTD level
  Arms: Phase Ib
Drug: afatinib — escalating dose
  Arms: Phase Ia, group 1

SUMMARY:
The aim of the study is to determine the Maximum Tolerated Dose (MTD) of afatinib in combination with 3-weekly trastuzumab in HER2 overexpressing cancer and to assess the efficacy of afatinib given at the MTD dosage, with 3-weekly trastuzumab in HER2 overexpressing metastatic breast cancer.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged 18 years and older
2. Patients with cancers overexpressing HER2 by Immunohistochemistry test( IHC) 3+ and/or IHC 2+ with positive gene amplification by FISH (confirmation on archived tissue needed)
3. Written informed consent that is consistent with ICH-GCP guidelines.
4. Patients must be eligible for treatment with trastuzumab.
5. Patients must have adequate organ function (kidney, liver, bone marrow, cardiac)
6. Eastern Cooperative Oncology Group (ECOG) = 0 or 1.
7. Measurable disease according to RECIST 1.1 (Phase Ib).

Exclusion criteria:

1. Active brain metastases.
2. Prior treatment with erbB family targeting therapies within the past four weeks before start of therapy or concomitantly with the trial other than trastuzumab and/or lapatinib.
3. Patients having more than 2 lines of chemotherapy for the treatment of metastatic breast cancer (Phase Ib).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-07-23 (Actual); Primary Completion 2016-06-23 (Actual); Study Completion 2016-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- France (3):
  - CTR Georges-François Leclerc, Dijon
  - CTR René Gauducheau, Saint-Herblain
  - INS Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HER2: Human Epidermal Growth Factor Receptor 2; RECIST,v1.1: Response Evaluation Criteria In Solid Tumors, version 1.1
Pre-assignment Details: Phase Ia: Open label, uncontrolled, dose escalation study of afatinib given continuously in combination with trastuzumab administered every 3 weeks. Phase Ib: Open label, uncontrolled study to explore the efficacy, safety, pharmacokinetics & biomarkers of afatinib at the MTD dosage, with 3- weekly trastuzumab.
Groups:
- Phase Ia: Afatinib 20mg+Trastuzumab 8 mg/kg: In each 21 day treatment cycle, patients were administered orally 20 mg afatinib tablet from Day 2 continuous daily administration in combination with trastuzumab. An initial loading dose of trastuzumab 8 mg/kg was administered via intravenous infusion at Day1 Cycle1, followed by trastuzumab 6 mg/kg every 3 weeks. Trastuzumab intravenous infusion, 90 minutes, infusion duration could be reduced to 30 minutes if well tolerated.
- Phase Ia: Afatinib 30mg+Trastuzumab 8 mg/kg: In each 21 day treatment cycle, patients were administered orally 30 mg afatinib tablet from Day 2 continuous daily administration in combination with trastuzumab. An initial loading dose of trastuzumab 8 mg/kg was administered via intravenous infusion at Day1 Cycle1, followed by trastuzumab 6 mg/kg every 3 weeks. Trastuzumab intravenous infusion, 90 minutes, infusion duration could be reduced to 30 minutes if well tolerated.
Period: Overall Study
Arm/Group | Phase Ia: Afatinib 20mg+Trastuzumab 8 mg/kg | Phase Ia: Afatinib 30mg+Trastuzumab 8 mg/kg
Started | 6 | 7
Completed | 0 | 0
Not Completed | 6 | 7
Not completed — Progressive disease | 4 | 5
Not completed — Other Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other than stated above | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This patient set includes all patients who were documented to have taken at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ia: Afatinib 20mg+Trastuzumab 8 mg/kg | Phase Ia: Afatinib 30mg+Trastuzumab 8 mg/kg | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (3.7) | 48.4 (7.6) | 54.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: MTD of Afatinib in Combination With Trastuzumab Based on the Number of Patients With DLTs During the First Treatment Cycle (Afatinib).
Description: Maximum Tolerated Dose (MTD) of Afatinib in combination with trastuzumab based on the number of patients with dose limiting toxicity (DLT) during the first treatment cycle (Dose escalation part). The MTD was defined as the highest dose studied at which the incidence of a DLT was less than 17% (i.e. 1/6 patients) during the first cycle.
  One patient in the Afa30+Trast8 cohort developed tumour lysis syndrome during the first course of treatment and was therefore not evaluable for the primary endpoint.
Time Frame: First 21 days treatment cycle
Population: Treated set: This analysis set includes all patients who were documented to have taken at least one dose of study medication.
Measure: Number; unit: mg
Groups:
- Phase Ia: Afatinib +Trastuzumab 8 mg/kg: In each 21 day treatment cycle, patients were administered orally afatinib tablet from Day 2 continuous daily administration in combination with trastuzumab. An initial loading dose of trastuzumab 8 mg/kg was administered via intravenous infusion at Day1 Cycle1, followed by trastuzumab 6 mg/kg every 3 weeks. Trastuzumab intravenous infusion, 90 minutes, infusion duration could be reduced to 30 minutes if well tolerated.
Arm/Group | Phase Ia: Afatinib +Trastuzumab 8 mg/kg
Number analyzed (Participants) | 12
mg | 20

2. Primary Outcome: Dose Limiting Toxicities During cycle1
Description: Number of Patients With Dose Limiting Toxicity (DLT) occurring during Cycle 1 based on the investigator assessment.
  One patient in the Afa30+Trast8 cohort developed tumour lysis syndrome during the first course of treatment and was therefore not evaluable for the primary endpoint.
Time Frame: First 21-day treatment cycle
Population: Treated set
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ia: Afatinib 20mg+Trastuzumab 8 mg/kg | Phase Ia: Afatinib 30mg+Trastuzumab 8 mg/kg
Number analyzed (Participants) | 6 | 6
Participants | 1 | 2

3. Secondary Outcome: Best Overall Response (BOR)
Description: BOR represents the best response a patient had during their time in study from start of treatment until progression, the last evaluable assessment in absence of progression or start of subsequent anticancer therapy. For patients that died, BOR was to be calculated based on data up to last evaluable RECIST,v1.1 assessment prior to death. Death did not contribute as PD for BOR. As per RECIST v1.1 for target lesions (TL) & assessed by MRI: CR: Disappearance of all TL,all non-TL, & no new lesion. Any pathological lymph nodes must have had reduction in the short axis to <10 mm. PR: At least 30% decrease in sum of the longest diameter (SLD) of TL taking as reference the baseline SLD. PD: At least a 20% increase in SLD of TL taking as reference the smallest SLD recorded since treatment started, together with an absolute increase in SLD of at least 5mm. SD: Neither sufficient shrinkage to qualify for PR, taking as reference the baseline SLD, nor sufficient increase to qualify for PD.
Time Frame: Post baseline tumour-imaging was performed at every 6 weeks (in the week preceding the start of Cycles 3, 5, 7, 9, 11, etc.) until End of Treatment (EOT); up to 33 months
Population: Treated set
  Missing: First image time point not reached before discontinuation.
Measure: Number; unit: percentage of participants
Arm/Group | Phase Ia: Afatinib 20mg+Trastuzumab 8 mg/kg | Phase Ia: Afatinib 30mg+Trastuzumab 8 mg/kg
Number analyzed (Participants) | 6 | 7
percentage of participants
  Complete Response (CR) | 0.0 | 0.0
  Partial Response (PR) | 16.7 | 0.0
  Stable Disease (SD) | 16.7 | 100.0
  Progressive Disease (PD) | 50.0 | 0.0
  Missing | 16.7 | 0.0
  Not Evaluable | 0.0 | 0.0

4. Secondary Outcome: Objective Response
Description: Objective Response (OR) was defined as best overall response of complete response (CR) or partial response (PR), where best overall response was determined according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 from first administration of study medication until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy. As Per RECIST v1.1 for target lesions (TL) & assessed by MRI: CR: Disappearance of all TL,all non-TL, & no new lesion. Any pathological lymph nodes must have had reduction in the short axis to <10 mm. PR: At least 30% decrease in sum of the longest diameter (SLD) of TL taking as reference the baseline SLD.
Time Frame: Post baseline tumour-imaging was performed at every 6 weeks (in the week preceding the start of Cycles 3, 5, 7, 9, 11, etc.) until EOT; up to 33 months
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Phase Ia: Afatinib 20mg+Trastuzumab 8 mg/kg | Phase Ia: Afatinib 30mg+Trastuzumab 8 mg/kg
Number analyzed (Participants) | 6 | 7
percentage of participants | 16.7 | 0.0

5. Secondary Outcome: Clinical Benefit
Description: Clinical benefit was defined as best overall response of CR or PR or stable disease (SD) where best overall response is defined according to RECIST version 1.1 from first treatment administration until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy.
  As Per RECIST v1.1 for target lesions (TL) & assessed by MRI: CR: Disappearance of all TL,all non-TL, & no new lesion. Any pathological lymph nodes must have had reduction in the short axis to <10 mm. PR: At least 30% decrease in sum of the longest diameter (SLD) of TL taking as reference the baseline SLD. SD: Neither sufficient shrinkage to qualify for PR, taking as reference the baseline SLD, nor sufficient increase to qualify for PD.
Time Frame: as for outcome 4
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Phase Ia: Afatinib 20mg+Trastuzumab 8 mg/kg | Phase Ia: Afatinib 30mg+Trastuzumab 8 mg/kg
Number analyzed (Participants) | 6 | 7
percentage of participants | 33.3 | 100.0

ADVERSE EVENTS:
Time Frame: From first dose administration of the study medication to 28 days after last drug administration; up to 33 months
Arm/Group | Phase Ia: Afatinib 20mg+Trastuzumab 8 mg/kg | Phase Ia: Afatinib 30mg+Trastuzumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 4/6 | 4/7
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ia: Afatinib 20mg+Trastuzumab 8 mg/kg (N=6) | Phase Ia: Afatinib 30mg+Trastuzumab 8 mg/kg (N=7)
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ia: Afatinib 20mg+Trastuzumab 8 mg/kg (N=6) | Phase Ia: Afatinib 30mg+Trastuzumab 8 mg/kg (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiotoxicity (Cardiac disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 6
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Perianal erythema (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3
Tongue oedema (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 4 | 5
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Xerosis (General disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2
Conjunctivitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 1
Paronychia (Infections and infestations) | 1 | 5
Rash pustular (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 2
Glomerular filtration rate decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Phase Ib was not started due to the discontinuation of afatinib development in HER2 overexpressing metastatic breast cancer and also the availability of other approved efficacious treatment options.Thus the results are not provided for Phase Ib.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.